CLINICAL TRIAL: NCT03994887
Title: Interest of the Study of Electroencephalogram and Peripheral Vegetative Markers for the Evaluation of Nociception Under General Anesthesia.
Acronym: BRAIN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study not started
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18CH168; 2019-A00201-56 (Other: ANSM)
Record Dates: First submitted 2019-06-07; First posted 2019-06-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: General Anesthesia
Keywords: General anesthesia; Surgery; Free Head

STUDY DESIGN:
Intervention Model Description: This is a monocentric and prospective observational study on the physiology of nociception under general anesthesia. The patient will be his own witness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients under general anesthesia will be included.
  Interventions: Device: Experimental group

INTERVENTIONS:
Device: Experimental group — EEG acquisition system BioSemi (Amsterdam, the Netherlands), enabling real-time measurement and continuous recording of EEG on up to 128 leads.

SUMMARY:
General anesthesia (GA) is a state of loss of consciousness induced by anesthetic products. In a GA, two classes of products are usually used: on the one hand, hypnotics that are responsible for the sleep component (hypnosis) and memory loss (amnesia), and on the other hand opioids that have an analgesic role.

The doses of hypnotic and morphine necessary to achieve this state of loss of consciousness and lack of response to painful stimulation vary from subject to subject, and during surgery depending on the intensity of the stimulus, requiring permanent adaptation to avoid overdose or underdosing, responsible for morbidity.

Several monitors of the hypnotic component have been developed in recent years, which can now be used routinely, such as the Bispectral Index (BIS) or Spectral Entropy.

However, there is currently no clinically validated technique for monitoring pain or the effect of opioids in the operating room.

Spectral analysis of the electroencephalogram (EEG) revealed a significant decrease (-30%) in alpha spectral power, observed specifically in painful experimental conditions in healthy awake subjects. On the other hand, a painful experience is accompanied by transient changes in various parameters under vegetative control, whether cardiovascular, cutaneous or pupillary, essentially underpinned by the activation of the sympathetic system.

The investigators hypothesize that a real-time dynamic analysis of the spectral power of EEG combined with that of cardiovascular vegetative parameters, cutaneous conductance and pupillary diameter is likely to be a marker of nociception under GA.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security scheme
* Over 18 years old
* To be operated on a regulated surgery allowing access to the head and to one eye, under AG, in the operating theater of the CHU of Saint-Etienne
* And having given his free, informed, written and signed consent.

Exclusion Criteria:

* Subject to a measure of legal protection (tutelage, guardianship)
* Admitted for emergency surgery
* With known allergy to any of the anesthetic agents used in the study
* Having been asleep under general anesthesia in the 7 days preceding the intervention
* A pacemaker or heart transplant patient
* With a history of Parkinson's disease, insulin-dependent or non-insulin-dependent diabetes at a dysautonomic stage or chronic alcoholism at a dysautonomia stage
* With psychiatric history or severe depression
* Presenting a peripheral or central neurological pathology that may modify the physiological responses to nociceptive stimulation
* With abnormal heart rhythm (atrial fibrillation or frequent extrasystoles)
* Treated for arterial hypertension with angiotensin type 2 receptor antagonists
* Treated with anti-arrhythmic, α- or β-blocking, which would make the interpretation of the results more difficult
* With chronic pain
* Treated with morphine or long-term neuroleptic
* Consuming cannabis or another narcotic
* Presenting bilateral ocular pathology that may interfere with pupillary dilatation
* Or refusing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
ElectroEncephaloGram (EEG) Alpha spectral power | 1 day
  variations of the EEG parameters (spectral power of the alpha rhythms), during nociceptive stimuli performed under AG at constant hypnosis depth (BIS between 50 and 60), without and after injection of a standardized dose of morphine (0.2 μg / kg of sufentanil based on the theoretical weight) of the patient).

SECONDARY OUTCOMES:
Beta spectral power | 1 day
  variations of the EEG parameters (spectral power of the beta rhythms), during nociceptive stimuli performed under AG at constant hypnosis depth (BIS between 50 and 60), without and after injection of a standardized dose of morphine (0.2 μg / kg of sufentanil based on the theoretical weight) of the patient).
gamma spectral power | 1 day
  variations of the EEG parameters (spectral power of the gamma rhythms), during nociceptive stimuli performed under AG at constant hypnosis depth (BIS between 50 and 60), without and after injection of a standardized dose of morphine (0.2 μg / kg of sufentanil based on the theoretical weight) of the patient).
delta spectral power | 1 day
  variations of the EEG parameters (spectral power of the delta rhythms), during nociceptive stimuli performed under AG at constant hypnosis depth (BIS between 50 and 60), without and after injection of a standardized dose of morphine (0.2 μg / kg of sufentanil based on the theoretical weight) of the patient).
theta spectral power | 1 day
  variations of the EEG parameters (spectral power of the tetha rhythms), during nociceptive stimuli performed under AG at constant hypnosis depth (BIS between 50 and 60), without and after injection of a standardized dose of morphine (0.2 μg / kg of sufentanil based on the theoretical weight) of the patient).

OTHER OUTCOMES:
Low frequency spectral power | 1 day
  Low Frequence : 0,04-0,15 Hz on EEG in nociceptive stimuli performed under GA at constant hypnosis depth, without and after injection of a standardized dose of morphine (0.2 µg/kg sufentanil based on the patient's theoretical weight)
High frequency spectral power | 1 day
  High frequency (HF : 0,15-0,4 Hz) on EEG in nociceptive stimuli performed under GA at constant hypnosis depth, without and after injection of a standardized dose of morphine (0.2 µg/kg sufentanil based on the patient's theoretical weight)
Cutaneous conductance | 1 day
  The cutaneous conductance will be given by the Nociception Level index (NoL®)
Pupil dilation reflex | 1 day
  The pupillary dilation reflex will be given by the AlgiScan® videopupillometer.

CONTACTS AND LOCATIONS:
Overall Officials: DAVID CHARIER, MD, Principal Investigator — CHU DE ST ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No